CLINICAL TRIAL: NCT03200522
Title: Western Versus Prudent Diet Feeding Study in Adult Women With Asthma
Brief Title: BREATHE-Easy Trial
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding completion date passed, inadequate enrollment
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); University of Nebraska (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: IRB00111434; 4KL2TR001077-04 (NIH)
Record Dates: First submitted 2017-06-21; First posted 2017-06-27 (Actual); Last update posted 2021-09-14 (Actual); Status verified 2021-08

CONDITIONS: Asthma
Keywords: Asthma, Diet
MeSH Terms: conditions — Asthma | interventions — Diet, Healthy; Diet, Western

STUDY DESIGN:
Intervention Model Description: This is a randomized crossover pilot trial to evaluate the feasibility of a Western and prudent diet feeding study in Baltimore City adults with asthma.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Participants and nutrition staff will be aware of randomization assignments. All other study staff and the investigators will be blinded to assignment during the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prudent diet then Western diet (Active Comparator): Participants randomized to this arm will received 6 days of meals consistent with a Prudent diet, followed by a washout period, and then 6 days of meals consistent with a Western diet.
  Interventions: Other: Prudent diet; Other: Western diet
- Western diet then Prudent diet (Active Comparator): Participants randomized to this arm will received 6 days of meals consistent with a Western diet, followed by a washout period, and then 6 days of meals consistent with a Prudent diet.
  Interventions: Other: Prudent diet; Other: Western diet

INTERVENTIONS:
Other: Prudent diet — Six days of meals provided with high amounts of fruits and vegetables, whole grains, fiber, omega-3 fatty acids, low-fat dairy products, and overall high levels of antioxidants.
Other: Western diet — Six days of meals provided with high amounts of processed foods, fast foods, sweets, omega-6 fatty acids, and a low intake of fiber.

SUMMARY:
This research is being done to evaluate the feasibility of a prudent versus Western diet feeding study in women with asthma in Baltimore City. The results of this research will provide data to appropriately design a definitive study looking at the differential effects of these two diets on asthma health.

DETAILED DESCRIPTION:
The investigators are interested in the effects of two different diets on asthma health. The first, a prudent diet, consists of a high intake of fruits and vegetables, whole grains, fiber, omega-3 fatty acids, low-fat dairy products, and overall high levels of antioxidants (which may protect the lungs and the body against inflammation in patients with asthma). The second, a Western diet, consists of a high intake of processed foods, fast foods, sweets, omega-6 fatty acids, and a low intake of fiber (which may promote inflammation in the lungs and the body of patients with asthma).

This pilot study will test the feasibility/acceptability of the study design in providing these two diets to participants over a short period of time (6 days per diet), and gather preliminary data on asthma health outcomes that will be used to design a larger, definitive trial. Each participant will be randomly (by chance, like flipping a coin) assigned to start with one of these diets. All foods in each of the diets will be supplied by the study, and participants will be expected to eat all of the food provided and only the food provided for the next 6 days. The investigators will make sure that each participant gets enough food for what their body needs, based on a visit with a nutritionist at the beginning of the study. After eating either the Prudent diet or Western diet for 6 days, participants will have a 4-8 week break (or washout period), during which they will eat their usual diet. Then participants will begin the alternate dietary intervention (Prudent or Western) for another 6 days, depending on which they received first. Before and after each dietary period, researchers will ask questions, check lung function, and collect samples from participants to determine acceptability of the meals and study design, gather feedback on the intervention and overall study structure, assess for changes in lung health and asthma control, measure inflammation and oxidative stress in the lungs and systemic circulation, and evaluate changes in the airway and gut microbiome associated with the interventions that may influence the asthmatic response.

ELIGIBILITY:
Inclusion criteria:

* Age 18-55
* Female
* Obese (BMI>30kg/m2)
* Not breastfeeding
* Diagnosis of asthma, defined as

  * Physician diagnosis of asthma, and
  * Current treatment for asthma by a healthcare provider within the preceding twelve months. (Current asthma treatment defined as regular use of asthma medications. Asthma medications include short and long acting adrenergic bronchodilators, bronchodilator combinations, inhaled anticholinergics, inhaled corticosteroids, cromolyn sodium and nedocromil, leukotriene modifiers and methylxanthines.)
* Stable asthma, defined by no asthma exacerbation (ED visit, course of increased systemic steroids, or urgent health care visit for asthma) during the prior four weeks.
* Symptomatic asthma (Asthma Control Test <20 at baseline screening visit)
* Non-smoker, defined by no cigarettes in the past year and a negative urine cotinine
* No other major pulmonary disease such as cystic fibrosis or chronic obstructive pulmonary disease
* Willing to eat study diet and nothing else for each of the 6 days of controlled feeding

Exclusion criteria:

* Chronic oral steroid therapy (daily)
* Oral corticosteroid use within the past 4 weeks
* Respiratory tract infection within the past 4 weeks
* Significant medical issues such as heart disease or poorly controlled hypertension, type 1 diabetes, poorly controlled type 2 diabetes, or hypothyroidism that would interfere with collection of outcome measures or present safety issues in the opinion of the Principal Investigator
* Pregnancy (self-report), planning a pregnancy, or nursing/breastfeeding mothers
* Food allergy that interferes with ability to complete the study
* Food preferences, intolerances, or dietary requirements that would interfere with diet adherence
* Taking vitamin supplements
* Planned dietary changes during the study period
* Use of coumadin
* Consumption of more than 14 alcoholic drinks per week, or consumption of 6 or more drinks on an occasion, one or more occasions per week
* Forced expiratory volume at one second (FEV1)<1.5 liters or <60% predicted
* Inability to perform acceptable spirometry
* Any condition or compliance issue which in the opinion of the investigator might interfere with participation in the study
* Lack of appropriate food refrigeration and preparation equipment (oven or microwave)
* Inability to produce adequate sputum following induction with hypertonic saline neb

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 3 (Actual)
Dates: Start 2017-10-12 (Actual); Primary Completion 2018-07-03 (Actual); Study Completion 2018-07-03 (Actual)

PRIMARY OUTCOMES:
Feasibility: participant feedback | At conclusion of second feeding period, 7-14 weeks post-enrollment
  We will measure this via questionnaire at the final study visit.
Feasibility: adherence to diet | Completed daily during each of the two, 6-day feeding periods.
  Daily adherence diaries completed by each participant during each dietary intervention.
Feasibility: serum carotenoids | Difference between day 1 and day 7 of each feeding period
  Serum carotenoids will be measured the morning prior to initiating each feeding period and the morning following completion of each 6-day feeding period.
Feasibility: serum lipids | Difference between day 1 and day 7 of each feeding period
  Serum lipids will be measured the morning prior to initiating each feeding period and the morning following completion of each 6-day feeding period.
Feasibility: serum free fatty acids | Difference between day 1 and day 7 of each feeding period
  Serum free fatty acids will be measured the morning prior to initiating each feeding period and the morning following completion of each 6-day feeding period.
Feasibility: obtaining sputum samples | Difference between baseline levels and levels on day 7 of each feeding period.
  Induced sputum will be collected for analysis of airway inflammation, a proposed key outcome for a definitive future trial.

SECONDARY OUTCOMES:
Asthma Quality of Life Questionnaire (AQLQ) | Difference between baseline levels and levels on day 7 of each feeding period.
  Asthma Quality of Life Questionnaire (AQLQ) is a 32 item questionnaire and each question uses a 7-point Likert scale (7 = not impaired at all - 1 = severely impaired).
Asthma Symptom Utility Index (ASUI) | Difference between day 1 and day 7 of each feeding period
  Asthma Symptom Utility Index (ASUI, range 0-1, higher score denoting fewer symptoms) will be measured.
Asthma Control Test (ACT) | Difference between baseline levels and levels on day 7 of each feeding period.
  Asthma Control Test (ACT, range 5-25, higher score denoting better asthma control).
Daily symptoms | Completed daily during each of the two, 6-day feeding periods.
  Daily symptom diaries completed by each participant during each dietary intervention.
FEV1 | Difference between day 1 and day 7 of each feeding period
  Spirometry will be measured according to the American Thoracic Society standards. The forced expiratory volume in one second (FEV1) will be assessed.
FVC | Difference between day 1 and day 7 of each feeding period
  Spirometry will be measured according to the American Thoracic Society standards. The forced vital capacity (FVC) will be assessed.
FEV1/FVC ratio | Difference between day 1 and day 7 of each feeding period
  Spirometry will be measured according to the American Thoracic Society standards. The forced expiratory volume in one second (FEV1)/forced vital capacity (FVC) ratio will be assessed.
Albuterol inhaler (rescue medication) use | Completed daily during each of the two, 6-day feeding periods.
  Daily diaries of self-reported albuterol use completed by each participant during each dietary intervention.
Exhaled nitric oxide | Difference between day 1 and day 7 of each feeding period.
  Exhaled nitric oxide is an indicator of airway inflammation and will be measured according to American Thoracic Society standards.
Markers of systemic Th2 inflammation | Difference between day 1 and day 7 of each feeding period.
  Serum and urine will be assessed for markers of Th2 inflammation.
Markers of airway Th2 inflammation | Difference between baseline levels and levels on day 7 of each feeding period.
  Sputum will be assessed for markers of Th2 inflammation.
Markers of systemic Th1 inflammation | Difference between day 1 and day 7 of each feeding period.
  Serum will be assessed for markers of Th1 inflammation.
Markers of airway Th1 inflammation | Difference between baseline levels and levels on day 7 of each feeding period.
  Sputum will be assessed for markers of Th1 inflammation.
Markers of systemic oxidative stress | Difference between day 1 and day 7 of each feeding period.
  Serum and urine will be assessed for markers of oxidative stress.
Markers of airway oxidative stress | Difference between baseline levels and levels on day 7 of each feeding period.
  Sputum will be assessed for markers of oxidative stress.
Upper airway microbiome | Difference between microbial community composition on day 1 and day 7 of each feeding period.
  Microbiome assessment via nasal swab collection.
Lower airway microbiome | Difference in microbial community composition between baseline and day 7 of each feeding period.
  Microbiome assessment via sputum collection.
Gut microbiome | Difference between microbial community composition on day 1 and day 7 of each feeding period.
  Microbiome assessment via stool collection.

CONTACTS AND LOCATIONS:
Overall Officials: Emily Brigham, MD, MHS, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-08-10): https://cdn.clinicaltrials.gov/large-docs/22/NCT03200522/Prot_SAP_000.pdf